CLINICAL TRIAL: NCT06622096
Title: Rationalization of Laboratory Tests in the ICU: Current State of Play
Brief Title: Evaluation of Lab Exams Accuracy in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, head of the ICU department, Mongi Slim Hospital
Other Study IDs: Lab exams in the ICU
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Laboratory Testing; Intensive Care Unit ICU; Accuracy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICU patients with a predicted length of stay > 24 hours
  Interventions: Diagnostic Test: Evaluation of laboratory exams prescription

INTERVENTIONS:
Diagnostic Test: Evaluation of laboratory exams prescription — Evaluation of laboratory exams prescription

SUMMARY:
prospective, observational descriptive study assessing the accuracy of laboratory exams in the ICU.

DETAILED DESCRIPTION:
Laboratory exams prescription for ICU patients was evaluated daily and their accuracy was determined according to locally implemented prescription protocol and to their abnormalities and the impact on further therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* All adults ICU patients with a length of stay>24 hours

Exclusion Criteria:

* Patients transferred from other ICUs
* Currently unavailable laboratory tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted in the ICU for more than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Blood loss due to laboratory tests | 7 days
  evolution of hemoglobin levels before and after laboratory tests

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim University Hospital, Tunis, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No